CLINICAL TRIAL: NCT05052788
Title: Optical Coherence Tomography Angiography in Patients With Cerebral Small Vessel Disease.
Brief Title: OCT Angio in Cerebral Small Vessel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: 930107130
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Small Vessel Disease and OCT Angio
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: 40 patients according to inclusion criteria .
  Interventions: Device: Optical coherence tomography angiography
- Control group: 20 normal people with no history of previous brain insult and with free neurological examination .
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Device: Optical coherence tomography angiography — OCT-A detects the motion of blood using intrinsic signals to capture the location of blood vessels. Despite its insensitivity to leakage and the relatively small field of view, the development of OCT-A has the potential to improve our knowledge of the physiology and pathophysiology of the eye.
  MRI as a stroke protocol, including T1 and T2 weighted images, diffusion weighted images (DWI), fluid attenuated inversion recovery (FLAIR), magnetic resonance angiography (MRA), and gradient recalled echo (GRE) T2* weighted images, using a machine 1.5 tesla General Electric machine .
  Other Names: MRI

SUMMARY:
The aim of the study is to: - detect changes in retinal structure and microvasculature in patients with cerebral small vessel disease using optical coherence tomography angiography , correlate these changes with brain imaging markers and determine if ( OCTA ) can be used as a screening tool for cerebral small vessel disease.

DETAILED DESCRIPTION:
Cerebral small vessel disease ( CSVD ) refers to all pathological changes affecting the small vasculature of the brain including; small perforating arterioles,capillaries and venules.

Vascular risk factors that are commonly found in large vessel disease have shown to contribute to CSVD, as well, including hypertension, diabetes mellitus, smoking and dyslipidemia.Also old age is considered to be a risk factor as the prevelance of CSVD increases with age affecting nearly 5 % of people aged 50 years and almost 100% in those older than 90 years .

Cerebral amyloid angiopathy is one of the suggested underlying pathologies in some cases of CSVD.

Clinically, CSVD accounts for 25% of ischemic strokes and 50% of dementias . It may present as acute events (focal neurological deficit ) known as lacunar syndrome or chronic events as mild cognitive dysfunction, dementia, mood disorders, gait disturbance, sleep disorder and urinary incontinence. Also, it may be a symptomatic.

Although CSVD is a common reason for strokes and vascular dementia, pathogenesis is still poorly understood . It is suggested that the endothelial dysfunction in cerebral microvessels may be a key problem. Endothelial failure leads to increased permeability and increased leakage into the vessel wall and the surrounding tissue , damaging of the vessel wall , inflammation, demyelination, glial scar formation , thickening and stiffness of vessels leading to failure of autoregulation, narrowing of the lumen and occlusion , causing featured focal ischemic lesions in the brain parenchyma.

Neuroimaging markers seen on MRI are classified into: Recent small subcortical infarct (DWI), Lacune of presumed vascular origin (FLAIR), White matter hyperintensity of presumed vascular origin (FLAIR), Perivascular space (T1 , T2), cerebral microbleed (T2*-weighted GRE/SWI).

The changes in brain microvasculature are difficult to be visualized in vivo . Because of similarities between brain and retina in anatomy , embryology and physiology , investigating the retinal vessels network may reflect the brain condition.

Optical coherence tomography angiography ( OCTA ) is a novel, real-time and noninvasive technique to detect retinal and choroidal blood flow in vivo.

The retinal capillary network is arranged anatomically into several layers as following ; 3 macular plexuses, 4 plexuses in peripapillary region and one capillary layer in midequatorial and anterior zones where the retina is thinner. OCTA devices are based on (en face) approach to get information of the superficial and deep plexuses. 4 en face zones are detected ; superfacial plexus in ganglion cell layer, deep plexus, photoreceptors(outer retina) and choroiocapillaries. For each en face zone , the indices of perfusion could be reached.

OCTA has a big advantage over classic methods as retinal microvasculature are segmented into layers and can be visualized and quantified more accurately . It is a safe and rapid technique giving a vascular map of retinal blood flow without using intravenous dye.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed clinically with small vessel disease and verified by MRI.
2. must be at age of 50 or more.

Exclusion Criteria:

1. large vessel disease or non-ischemic leukoencephalopathy.
2. Patients with any type of cerebral haemorrhage .
3. Diabetic patients .
4. concurrent retinal diseases as epiretinal memberane and macular degeneration.
5. Past history of retinal operation or ocular surgery except for cataract surgery.
6. An history of glaucoma or optic neuropathy.
7. hematological diseases and coagulopathies.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of people, patients (case group) and (control group), both groups are frequency matched in age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of retinal microvasculature changes using OCT angio (OCTA). | Anticipated 2 months
  OCTA can detect five parameters:
  ( macular vessel density, macular thickness, ganglion cell layer thickness, pericapillary nerve fiber layer thickness and pericapillary vessel density ).
  Compare between case and control group using OCTA parameters then correlate OCTA parameters with clinical and neurological imaging parameters.

REFERENCES:
- [Background] Cannistraro RJ, Badi M, Eidelman BH, Dickson DW, Middlebrooks EH, Meschia JF. CNS small vessel disease: A clinical review. Neurology. 2019 Jun 11;92(24):1146-1156. doi: 10.1212/WNL.0000000000007654. Epub 2019 May 29. PMID 31142635
- [Background] Chen X, Wang J, Shan Y, Cai W, Liu S, Hu M, Liao S, Huang X, Zhang B, Wang Y, Lu Z. Cerebral small vessel disease: neuroimaging markers and clinical implication. J Neurol. 2019 Oct;266(10):2347-2362. doi: 10.1007/s00415-018-9077-3. Epub 2018 Oct 5. PMID 30291424